CLINICAL TRIAL: NCT02580071
Title: An Open Label, Non-randomized, Clinical Study of Chinese Medicine, Sheng-Yu-Tang, for Immune Reconstitution Following Peripheral Blood Stem Cell Transplantation in >CR1 (Complete Remission) and Refractory Acute Leukemia Patients
Brief Title: Chinese Herbal Medicine for Immune Reconstitution Following HSCT in Acute Leukemia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Hung-Rong Yen, Dr. Hung-Rong Yen, MD, PhD, China Medical University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CMUH104-REC3-066
Record Dates: First submitted 2015-10-16; First posted 2015-10-20 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Acute Leukemia
Keywords: Hematopoietic Stem Cell Transplant; Chinese Herbal Medicine; immune reconstitution; clinical trial; ALL; AML

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sheng-Yu-Tang (Experimental): Treatment group will receive standard of care, as well as:
  2-3 months post-HSCT, patients will be administered the herbal formula Sheng-Yu-Tang (聖愈湯), which they will receive for 6 months. The herbal formula will be provided from a GMP herbal company and will be given in granulated form.
  Interventions: Dietary Supplement: Sheng-Yu-Tang
- Control (No Intervention): Control group will receive standard of care

INTERVENTIONS:
Dietary Supplement: Sheng-Yu-Tang — Granulated formula will be prescribed by KO DA Pharmaceutical co., LTD (科達) composition of formula is as follows: Radix Rehmanniae Praeparata 4g Radix Paeoniae Alba 4g Radix Astragali 4g Radix Ginseng 4g Radix Angelice Sinensis 2g Rhizoma Chuanxiong 2g (for preperation method and concentration ratio's please refer to manufacturers information)
  patients will be required to take 4.2gr, t.i.d (total of 12.6gr per day)
  Other Names: 聖愈湯; "Sagacious Cure Decoction"
  Arms: Sheng-Yu-Tang

SUMMARY:
The treatment options for high-risk acute leukemia patients are limited and these patients are often opt for hematopoietic stem cell transplant (HSCT). However studies show that prognosis following this last-resort therapy is bleak. At times, less than 70% of post-HSCT relapsed AML and ALL patients even achieve complete remission; median overall survival of these cohorts might not reach one year; and 3-year post-HSCT survival rates might be less than 20%.

The investigators plan to recruit acute leukemia patients from CMUH which are planned to receive HSCT, and follow the rate and quality of their immune reconstitution. As intervention, part of the patients will receive a Chinese medicine herbal formula, which they will take for 6 months.Differences between the 1-year post-HSCT condition of patients will be examined.

DETAILED DESCRIPTION:
We hope to enroll 50 high-risk acute leukemia patients after receiving HSCT at China Medical University Hospital. Thereupon, patients will be consecutively recruited to treatment group (25 patients) where they will be prescribed Sheng Yu Tang (聖愈湯, SYT) 2 months following HSCT, for a period of 6 months, in conjunction with the standard-care treatment. We predict that not all patients will be interested in taking SYT, patients which are not interested in entering treatment group will be offered to join a control group (25 patients) which will receive standard-care treatment.

Since HSCT patients go through routine blood examinations, this study will request to extract a further 20ml of peripheral blood once a month and an additional 20ml of bone marrow at beginning of HSCT and the following routine aspirations (est.:0, +3, +6, +9, +12 month). Both treatment and control group will be required to contribute peripheral blood and bone marrow sample.Blood samples will be collected until patients reach 1-year post-HSCT, and flow cytometry will be used to examine the difference in immune reconstitution rate between the two groups. As secondary outcome measurements, this study will make use of the minimal residual disease (MRD) measured, frequency of opportunistic infections, hospitalizations and results of other routine check-up which recorded in patient history.

ELIGIBILITY:
Inclusion Criteria:

* Discharged from hospital.
* Diagnosed with ALL, AML or MDS-AML.
* Received allogeneic or haploidentical peripheral blood HSCT.
* Willing to supply blood samples for analysis.
* Willing to comply with all study interventions and follow-ups.

Exclusion Criteria:

* unable, due to known allergy or any other reason, to orally take Chinese Herbal Medicine.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-10; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Peripheral blood Immune reconstitution | 1 year

SECONDARY OUTCOMES:
Minimal residual disease (MRD) | 1 year
Bone marrow Immune reconstitution | 1 year
complete blood count | 1 year
  WBC count WBC differential RBC count Hematocrit Hemoglobin Platelet Mean platelet volume ALT/AST gamma gt
opportunistic infection | 1 year
  Aspergillus Candida Herpes simplex virus (HSV) Cytomegalovirus (CMV) Varicella-zoster virus (VZV) Human herpes virus 6 (HHV6) Epstein-Barr virus
GvHD | 1 year
frequency of hospitalizations | 1 year
Quality of Life | 1 year
  QLQ-C30 Chinese Mandarin

OTHER OUTCOMES:
Wang Q. constitution in Chinese medicine questionnaire | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Rong Yen, M.D., Ph.D., Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

REFERENCES:
- [Derived] Fleischer T, Chang TT, Chiang JH, Yen HR. A Controlled Trial of Sheng-Yu-Tang for Post-Hematopoietic Stem Cell Transplantation Leukemia Patients: A Proposed Protocol and Insights From a Preliminary Pilot Study. Integr Cancer Ther. 2018 Sep;17(3):665-673. doi: 10.1177/1534735418756736. Epub 2018 Feb 11. PMID 29431027